CLINICAL TRIAL: NCT03631368
Title: Treatment of Hypertrophic Scars With Intradermal Botox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Roy G. Geronemus, M.D. (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor-Investigator, Roy G. Geronemus, M.D., Principal Investigator, Laser and Skin Surgery Center of New York
Organization: Laser and Skin Surgery Center of New York (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSSC-BOTOXSCAR-2018
Record Dates: First submitted 2018-08-09; First posted 2018-08-15 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Hypertrophic Scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Botox (Experimental)
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — Intradermal injection with Botox 100U/mL will be performed using a 25g needle. Each subject will receive three treatments spaced 1 month apart.

SUMMARY:
This is a prospective, open label, single center, self-controlled clinical study to demonstrate the safety and efficacy of intradermal botulinum toxin in treating hypertrophic scarring.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female and male subjects between the ages 18-75.
2. Non-Smoker.
3. Fitzpatrick skin type I-VI.
4. Desire to improve hypertrophic scarring.
5. Able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Able to understand and provide written Informed Consent.

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding.
2. Presence of any active systemic or local infections.
3. Presence of active local skin disease that may alter wound healing.
4. Known allergy to botulinum toxin.
5. History of smoking in past 10 years.
6. History of chronic drug or alcohol abuse.
7. Inability to understand the protocol or to give informed consent.
8. History of cosmetic treatments in the area to be treated, including injectable filler of any type within the past year; Botox in the treatment area within the past 6 months; ablative or non-ablative resurfacing/rejuvenation laser treatment or light treatment within the past 6 months, dermabrasion or deep peels within the past 6 months; surgery to the area within the past 6 months.
9. History of intralesional corticosteroids or any other injectable medication to the area within the last 3 months.
10. History of topical corticosteroids to the area within the past 4 weeks.
11. History of any musculoskeletal disease or any weakness in the area to be treated.
12. As per the investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of hypertrophic scars based on the Subject and Observer Scar Assessment Scale | change from baseline at 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Laser & Skin Surgery Center of New York, New York, New York, United States